CLINICAL TRIAL: NCT06109506
Title: Towards a Tailored Approach for Patients With Acute Diverticulitis and Abscess Formation. A Multicenter Cohort Analysis
Acronym: DivAbsc2023
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Collaborators: Azienda Ospedaliero Universitaria di Cagliari (Other)
Responsible Party: Principal Investigator, Mauro Podda, Clinical Lecturer of Surgery, University of Cagliari
Other Study IDs: DivAbsc2023_1
Record Dates: First submitted 2023-10-23; First posted 2023-10-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Acute Diverticulitis; Diverticular Diseases; Diverticulitis of Sigmoid; Acute Diverticular Perforation; Diverticulitis, Colonic; Sepsis
Keywords: Acute diverticulitis; Diverticular abscess; Conservative treatment
MeSH Terms: conditions — Diverticular Diseases; Diverticulitis, Colonic; Sepsis | interventions — Conservative Treatment; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with diverticular abscess classified as Hinchey 2b (Subgroup)
  Interventions: Procedure: Conservative treatment with antibiotics and eventual percutaneous image-guided drainage of the abscess
- Patients with diverticular abscess >5 cm (Subgroup)
  Interventions: Procedure: Conservative treatment with antibiotics and eventual percutaneous image-guided drainage of the abscess

INTERVENTIONS:
Procedure: Conservative treatment with antibiotics and eventual percutaneous image-guided drainage of the abscess — Patients with acute diverticulitis and abscess formation are commonly treated with a conservative approach that includes endovenous antibiotics and, for abscesses > 4-5 cm, percutaneous image-guided drainage.

SUMMARY:
It is estimated that approximately 15% to 20% of the subjects with sigmoid diverticulosis will develop acute diverticulitis, with diverticular abscess as the most common complication of sigmoid diverticulitis.

While cases with free perforations and diffuse peritonitis require emergency surgery, in cases with contained perforation and abscess formation, the approach is initially conservative. Due to its relative rarity, the treatment of diverticular abscess is not based on high-quality scientific evidence. Abscess size of 4-6 cm is generally accepted as reasonable cutoff determining the choice of treatment between antibiotic therapy and antibiotic therapy plus percutaneous drainage of the abscess.

A subgroup of patients will fail the conservative approach and require a surgical rescue strategy. However, the real incidence for conservative treatment failure after non-operative management of acute diverticulitis with abscess remain poorly understood, the knowledge of which could improve decision-making processes, treatment strategies, patient counseling, and even modify the planned treatment strategy in patients deemed at highest risk.

The early recognition of patients who show clinical signs of ongoing and worsening intra-abdominal sepsis due to perforation is important to ensure the success of this strategy. In the light of these, knowledge of risk predictors for failure is of utmost importance.

Owing the contrasting evidence summary, we set up a multicenter retrospective cohort study that merges the cases from twelve high-volume centers for emergency surgery in Italy to assess the short-term outcomes of initial non-surgical treatment strategies for AD with abscess formation (Hinchey Ib and II) in a large number of patients, and identify risk factors associated with adverse outcomes, to help facilitate appropriate patient selection and assess the optimal treatment strategy for this peculiar subgroup of patients.

The purpose of this study is to describe the incidence and risk factors for conservative treatment (antibiotics alone or antibiotics plus percutaneous drainage) failure after non-operative management of acute diverticulitis with abscess using a large multicenter patient series.

The present study is designed as a multicenter retrospective observational study conducted at twelve secondary and tertiary Italian teaching surgical centers on CT-diagnosed hemodynamically stable patients (≥18 years) with perforated acute diverticulitis with abscess (with or without extraluminal air) initially treated non-surgically.

The rate of failure of non-operative treatment for complicated acute diverticulitis patients with abscess formation and the risk factors of failure of the non-surgical treatment will be assessed.

Failure of the conservative treatment is defined as lack of clinical improvement in the general conditions of the patient during index hospital admission, requiring urgent surgery to treat intra-abdominal sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age) patients
2. Patients diagnosed with acute diverticulitis with radiological findings of contained perforation (modified Hinchey classification Ib and IIa/b).
3. Patients who are initially managed conservatively according to contemporary guidelines.

Exclusion Criteria:

1. Patients with perforated diverticulitis with peritonitis (Hinchey III or IV stages).
2. Patients with clinically assessed generalized peritonitis.
3. Patients diagnosed with colonic cancer mimicking acute diverticulitis with abscess.
4. Requirement for urgent or emergent surgery decided immediately following hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient cohort consists of adult (≥18 years of age) patients with a diagnosis of acute diverticulitis complicated by localized intra-abdominal abscess formation with pericolic or pelvic localization and/or localized pericolic extraluminal air, corresponding to the modified Hinchey classification Ib and IIa/b. These patients should be managed conservatively according to contemporary guidelines, but still have a high probability for failure of conservative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with failure of the conservative treatment. | 15 days after the beginning of conservative treatment.
  Failure of the conservative treatment is defined as the need for emergency surgical therapy performed during the index hospitalization due to clinical deterioration in spite of initial diverticular abscess treatment with antibiotics +/- percutaneous drainage.

SECONDARY OUTCOMES:
Number of patients with recurrence of acute diverticulitis. | 90 days after initial successful conservative treatment and hospital discharge.
  Recurrence of symptomatic acute diverticulitis requiring a new hospital admission.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari Hospital, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Podda M, Ceresoli M, Di Martino M, Ortenzi M, Pellino G, Pata F, Ielpo B, Murzi V, Balla A, Lepiane P, Tamini N, De Carlo G, Davolio A, Di Saverio S, Cardinali L, Botteri E, Vettoretto N, Gelera PP, De Simone B, Grasso A, Clementi M, Meloni D, Poillucci G, Favi F, Rizzo R, Montori G, Procida G, Recchia I, Agresta F, Virdis F, Cioffi SPB, Pellegrini M, Sartelli M, Coccolini F, Catena F, Pisanu A. Towards a tailored approach for patients with acute diverticulitis and abscess formation. The DivAbsc2023 multicentre case-control study. Surg Endosc. 2024 Jun;38(6):3180-3194. doi: 10.1007/s00464-024-10793-z. Epub 2024 Apr 17. PMID 38632117